CLINICAL TRIAL: NCT04914520
Title: A Phase 1 Study to Assess the Safety, Tolerability, and Immunogenicity of VN-0200 After Intramuscular Injections in Japanese Healthy Adults and Elderly Subjects
Brief Title: Study of VN-0200 in Japanese Healthy Adults and Elderly Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: VN0200-A-J101; jRCT2031210069 (Other: Japan Registry of Clinical Trials)
Record Dates: First submitted 2021-05-19; First posted 2021-06-04 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-12

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: Respiratory Syncytial Virus Infections; VN0200
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Step 1: VN-0200 low dose (Experimental): Healthy adults subjects will be randomized to receive intramuscular injection of low dose of VAGA-9001a adjuvanted with low dose of MABH-9002b.
  Interventions: Biological: VN-0200
- Step 1: VN-0200 medium dose (Experimental): Healthy adults subjects will be randomized to receive intramuscular injection of medium dose of VAGA-9001a adjuvanted with medium dose of MABH-9002b.
  Interventions: Biological: VN-0200
- Step 1: VN-0200 high dose (Experimental): Healthy adults subjects will be randomized to receive intramuscular injection of high dose of VAGA-9001a adjuvanted with high dose of MABH-9002b.
  Interventions: Biological: VN-0200
- Step 1: Placebo (Placebo Comparator): Healthy adults and elderly subjects will be randomized to receive intramuscular injection of placebo.
  Interventions: Biological: Placebo
- Step 2: VN-0200 low dose (Experimental): Healthy elderly subjects will be randomized to receive intramuscular injection of low dose of VAGA-9001a adjuvanted with low dose of MABH-9002b.
  Interventions: Biological: VN-0200
- Step 2: VN-0200 dose medium dose (Experimental): Healthy elderly subjects will be randomized to receive intramuscular injection of medium dose of VAGA-9001a adjuvanted with medium dose of MABH-9002b.
  Interventions: Biological: VN-0200
- Step 2: VN-0200 high dose (Experimental): Healthy elderly subjects will be randomized to receive intramuscular injection of high dose of VAGA-9001a adjuvanted with high dose of MABH-9002b.
  Interventions: Biological: VN-0200
- Step 2: Placebo (Placebo Comparator): Healthy adults and elderly subjects will be randomized to receive intramuscular injection of placebo.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: VN-0200 — VN-0200 (antigen: VAGA-9001a, adjuvant: MABH-9002b) administered as an intramuscular injection into the deltoid muscle of the upper arm; 2 injections total
  Arms: Step 1: VN-0200 high dose; Step 1: VN-0200 low dose; Step 1: VN-0200 medium dose; Step 2: VN-0200 dose medium dose; Step 2: VN-0200 high dose; Step 2: VN-0200 low dose
Biological: Placebo — Placebo administered as an intramuscular injection into the deltoid muscle of the upper arm; 2 injections total
  Arms: Step 1: Placebo; Step 2: Placebo

SUMMARY:
This study will assess the safety, tolerability, and immunogenicity of VN-0200 after intramuscular injections in Japanese healthy adults and elderly subjects.

ELIGIBILITY:
Inclusion Criteria:

* Japanese
* Healthy adults aged ≥20 and ≤50 years (Step 1) or healthy elderly aged ≥65 and ≤80 years (at the time of informed consent)
* Body mass index (BMI) is ≥18.0 and <30.0 kg/m^2 (at screening)

Exclusion Criteria:

* Participants with a history of anaphylaxis or severe allergies due to food, medicine, insect bites, cosmetics, or vaccination
* Having alcohol or drug dependence, etc.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-06-11 (Actual); Primary Completion 2021-12-16 (Actual); Study Completion 2021-12-16 (Actual)

PRIMARY OUTCOMES:
Number of Participants Reporting Treatment-emergent Adverse Events | From first administration through 28 days post second administration
Number of Participants Reporting Local and Systemic Adverse Events | From first administration up to 14 days after second administration
Number of Participants Reporting Serious Adverse Events | From date of informed consent up to approximately 3 months

SECONDARY OUTCOMES:
Geometric Mean Fold Rise (GMFR) of Anti-RSV Specific Neutralizing Activity | Day 29 and Day 57 post-dose and at the time of discontinuation (whichever occurs first), up to approximately 2 months
Geometric Mean Titer (GMT) of Anti-VAGA-9001a IgG | Day 1 (pre-dose), Day 29 and Day 57 post-dose, and at the time of discontinuation (whichever occurs first), up to approximately 2 months
Geometric Mean Titer (GMT) of Anti-RSV IgG | Day 1 (pre-dose), Day 29 and Day 57 post-dose, and at the time of discontinuation (whichever occurs first), up to approximately 2 months
Number of IFN-γ spot-forming cells in PBMC Detected by ELISPOT | Day 1 (pre-dose), Day 29 and Day 57 post-dose, and at the time of discontinuation (whichever occurs first), up to approximately 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Leader, Study Director — Daiichi Sankyo
Locations (1):
- Medical Corporation Association Shinanokai Shinanozaka Clinic, Shinjuku-Ku, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No